CLINICAL TRIAL: NCT02281422
Title: An Open-label, Single-dose, Single-centre Study, Investigating the Pharmacokinetics of BIA 2-093 in Subjects With Various Degrees of Renal Impairment
Brief Title: An Open-label, Single-dose, Single-centre Study, Investigating the Pharmacokinetics of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-112
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 normal renal function (Other): normal renal function (creatinine clearance > 80 mL/min)
  Interventions: Drug: BIA 2-093
- Group 2 mild renal impairment (Other): mild renal impairment (creatinine clearance 50-80 mL/min)
  Interventions: Drug: BIA 2-093
- Group 3 moderate renal impairment (Other): moderate renal impairment (creatinine clearance 30-50 mL/min)
  Interventions: Drug: BIA 2-093
- Group 4 severe renal impairment (Other): severe renal impairment (creatinine clearance <30 mL/min)
  Interventions: Drug: BIA 2-093
- Group 5 end stage renal disease (Other): end stage renal disease, requiring haemodialysis (ESRD)
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093

SUMMARY:
Open-label, single-dose (BIA 2-093 800 mg tablet), single-centre study in five groups of subjects with various degrees of renal function based on creatinine clearance

DETAILED DESCRIPTION:
This was an open-label, single-dose (BIA 2-093 800 mg tablet), single-centre study in five groups of subjects with various degrees of renal function based on creatinine clearance (stages of renal function according to the Food and Drug Administration and the European Agency for the Evaluation of Medicinal Products Guidelines) for the evaluation of pharmacokinetics in patients with impaired renal function.

The trial commenced with Groups 1 and 2. An interim safety evaluation was conducted and, as there were no safety concerns, the trial continued with Groups 3 and 4. After another interim safety evaluation with the data from Groups 3 and 4, the trial commenced with Group 5.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age, with body mass not less than 50 kg.
* Female subjects had to be post-menopausal, surgically sterilized or using a reliable method of contraception.
* Subjects suffering from a chronic illness, other than hepatic impairment, had to have a stable condition, regarded by the investigator as unlikely to influence the outcome of the study.
* Renal failure, the extent of which, as measured by the creatinine clearance, resulted in recruitment to one of five renal function groups.
* Medical records indicating a stable serum creatinine (variation of not more than 30%), for at least 3 months prior to the screening visit (Groups 2 to 4 only), as determined by the clinical investigator. The sérum creatinine had to be stable to allow for an accurate determination of the creatinine clearance and therefore allowed for correct allocation to one of the renal function groups. Subjects who were recruited into Group 1 had normal renal function.

Exclusion Criteria:

* The receipt of any investigational drug within 30 days prior to this study.
* Clinically significant abnormal findings (as judged by the investigator) for the following parameters, except those consistent with findings in renal failure: haematology, biochemistry, clotting profile, urinalysis, vital signs or ECG screening tests.
* A history or laboratory evidence of hepatic impairment and/or disease. Owing to the metabolic pathway of BIA 2-093, any degree of hepatic impairment would have had a confounding effect on the PK analysis.
* Positive test for HIV-1 or HIV-2 Antibodies, Hepatitis B surface antigen and Hepatitis C Antibodies.

HIV positive patients, and patients with Hepatitis B and C, generally have a below average, and in some cases a markedly decreased, level of health owing to the nature of the respective infections and the natural course of the diseases, both of which are often complicated by an array of opportunistic illnesses. Their ill health would have been further worsened by the fact that the patients are invarious degrees of renal failure, which has its own, often debilitating, complications. If patients with HIV or Hepatitis B or C were included in the study, this could have led to statistical confusion when assessing the safety and tolerability parameters. This is because events reported by the patients, which may be a part of the spectrum of complaints in HIV positive patients and Hepatitis B and C patients, would have confounded the safety and tolerability analysis. Furthermore, Hepatitis B and C, which may cause an element of hepatic impairment, would have confounded the PK analysis due to the metabolic pathway of BIA 2-093. In addition, by administering the study medication to these subjects, any adverse events that might have occurred would have added to the discomfort of the patient.

* A history of any illness that, in the opinion of the Investigator and/or Sponsor, might have confounded the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Farmovs-Parexel, Bloemfontein, Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Normal Renal Function: normal renal function (creatinine clearance > 80 mL/min)
  BIA 2-093
- Group 2 Mild Renal Impairment: mild renal impairment (creatinine clearance 50-80 mL/min)
  BIA 2-093
- Group 3 Moderate Renal Impairment: moderate renal impairment (creatinine clearance 30-50 mL/min)
  BIA 2-093
- Group 4 Severe Renal Impairment: severe renal impairment (creatinine clearance <30 mL/min)
  BIA 2-093
- Group 5 End Stage Renal Disease: end stage renal disease, requiring haemodialysis (ESRD)
  BIA 2-093
Period: Overall Study
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease
Started | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 7 | 8 | 8 | 38
  >=65 years | 0 | 1 | 1 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 2 | 1 | 3 | 14
  Male | 7 | 1 | 6 | 7 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Peak Plasma Concentration
Description: BIA 2-194; BIA 2-195; Oxcarbazepine are BIA 2-093 metabolites
Time Frame: pre-dose and 1, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 5, 7, 9, 12, 24, 48, 72 and 96 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL
  Cmax (BIA 2-194) | 14286.790 (2988.340) | 18677.265 (4381.474) | 15055.632 (2513.170) | 14974.79 (4313.90) | 14510.197 (2149.176)
  Cmax (BIA 2-195) | 211.076 (61.0200) | 348.843 (69.739) | 410.828 (68.663) | 465.928 (201.988) | 359.798 (119.819)
  Cmax (Oxcarbazepine) | 138.339 (32.271) | 172.293 (43.431) | 157.629 (35.224) | 157.955 (61.354) | 208.473 (40.912)

2. Secondary Outcome: Tmax (hr) - Time at Which Cmax Occurred
Description: BIA 2-194; BIA 2-195; Oxcarbazepine are BIA 2-093 metabolites
  Cmax - maximum observed plasma drug concentration
Time Frame: pre-dose and 1, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 5, 7, 9, 12, 24, 48, 72 and 96 hours post-dose.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours
  Tmax (BIA 2-194) | 1.121 (0.530) | 1.327 (1.004) | 2.609 (2.504) | 2.680 (2.642) | 1.633 (1.069)
  Tmax (BIA 2-195) | 22.008 (4.2430) | 20.185 (5.557) | 26.172 (8.485) | 33.947 (12.824) | 10.773 (1.553)
  Tmax (Oxcarbazepine) | 2.396 (0.773) | 2.581 (0.681) | 3.970 (2.397) | 4.787 (3.172) | 4.260 (2.254)

3. Primary Outcome: AUC(0-12h) - AUC From Time Zero to 12h
Description: BIA 2-194; BIA 2-195; Oxcarbazepine are BIA 2-093 metabolites
  AUC - area under the plasma concentration versus time curve
Time Frame: pre-dose and 1, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 5, 7, 9, 12, 24, 48, 72 and 96 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng*h/mL
  AUC(0-12h) (BIA 2-194) | 105275.733 (21516.315) | 150945.034 (24049.320) | 138473.115 (19998.869) | 138262.814 (43286.475) | 134757.936 (18609.384)
  AUC(0-12h) (BIA 2-195) | 1522.370 (427.4400) | 2435.245 (681.175) | 2025.731 (419.930) | 2157.860 (1092.304) | 2690.584 (731.793)
  AUC(0-12h) (Oxcarbazepine) | 1218.276 (279.550) | 1388.146 (316.857) | 1460.113 (351.507) | 1496.463 (653.928) | 1832.298 (338.896)

ADVERSE EVENTS:
Arm/Group | Group 1 Normal Renal Function | Group 2 Mild Renal Impairment | Group 3 Moderate Renal Impairment | Group 4 Severe Renal Impairment | Group 5 End Stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 6/8 | 5/8 | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Normal Renal Function (N=8) | Group 2 Mild Renal Impairment (N=8) | Group 3 Moderate Renal Impairment (N=8) | Group 4 Severe Renal Impairment (N=8) | Group 5 End Stage Renal Disease (N=8)
HEADACHE (Nervous system disorders) | 5 | 3 | 2 | 1 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 3 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2 | 1 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
GENITAL PRURITUS FEMALE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other